CLINICAL TRIAL: NCT06929429
Title: Comparison of the Effects of Bilateral Sphenopalatine Ganglion and Infraorbital Nerve Blocks on Postoperative Recovery in Patients Undergoing Septorhinoplasty: A Prospective, Randomized, Double-Blind, Controlled Study"
Brief Title: Effect of Bilateral SPG and Infraorbital Nerve Blocks on Recovery After Septorhinoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Ömer Keklicek, MD, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/23
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Quality of Recovery (QoR-15); Sphenopalatine Ganglion Block; Infraorbital Nerve Block
Keywords: Septorhinoplasty; Quality of Recovery; Regional Anesthesia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups to receive either a bilateral sphenopalatine ganglion block or a bilateral infraorbital nerve block. Each participant will receive only one type of intervention, and the outcomes will be compared between the two groups.
Who Masked: Participant, Care Provider
Masking Description: The study is double-blinded. Neither the participants, the care providers, nor the outcome assessors are aware of group assignments. A separate staff member not involved in the study performs randomization and prepares the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sphenopalatine ganglion block (Active Comparator): Participants in this group will receive a bilateral sphenopalatine ganglion block using 4 mL of 0.5% bupivacaine via intranasal application after induction of general anesthesia and before the start of surgery.
  Interventions: Procedure: Bilateral Sphenopalatine Ganglion Block
- Infraorbital Nerve Block (Active Comparator): Participants in this group will receive a bilateral infraorbital nerve block with 4 mL of 0.5% bupivacaine administered under ultrasound guidance after induction of general anesthesia and before the start of surgery.
  Interventions: Procedure: Bilateral Infraorbital Nerve Block

INTERVENTIONS:
Procedure: Bilateral Sphenopalatine Ganglion Block — A bilateral sphenopalatine ganglion block will be performed after induction of general anesthesia using 4 mL of 0.5% bupivacaine. The local anesthetic will be applied intranasally with a cotton-tipped applicator placed parallel to the zygomatic arch and advanced to the posterior nasal cavity. The applicator will remain in place for 15 minutes.
  Arms: Sphenopalatine ganglion block
Procedure: Bilateral Infraorbital Nerve Block — A bilateral infraorbital nerve block will be performed after induction of general anesthesia using 4 mL of 0.5% bupivacaine per side. The block will be guided by linear ultrasound to identify the infraorbital foramen and administered with a 22G needle around the nerve. A 15-minute absorption period will be allowed before the surgical procedure begins.
  Arms: Infraorbital Nerve Block

SUMMARY:
This prospective, randomized, double-blind controlled study aims to compare the effects of bilateral sphenopalatine ganglion and infraorbital nerve blocks on postoperative recovery quality in patients undergoing elective septorhinoplasty under general anesthesia. A total of 90 adult patients (aged 18-65, ASA I-II) will be randomly assigned into two groups: Group 1 will receive bilateral sphenopalatine ganglion block, and Group 2 will receive bilateral infraorbital nerve block. Both blocks will be performed using 4 mL of 0.5% bupivacaine.

The primary outcome is the quality of recovery assessed 24 hours after surgery using the QoR-15 questionnaire. Secondary outcomes include intraoperative anesthetic consumption (propofol, remifentanil), emergence agitation (RASS scale), postoperative pain (VAS), need for rescue analgesics (morphine), postoperative nausea and vomiting (VDS), antiemetic consumption (ondansetron), facial edema and hematoma, and length of stay in the post-anesthesia care unit (PACU).

All procedures will follow standardized general anesthesia protocols. The study aims to determine which block technique provides superior postoperative recovery, better pain control, fewer side effects, and higher patient satisfaction. No placebo will be used, and no biological samples will be collected.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, controlled clinical trial designed to evaluate the effects of two regional anesthesia techniques-bilateral sphenopalatine ganglion block and bilateral infraorbital nerve block-on postoperative recovery quality in adult patients undergoing elective septorhinoplasty under general anesthesia.

A total of 90 patients aged 18-65 years, classified as ASA physical status I-II, will be randomly assigned into two groups using sealed opaque envelope randomization by a non-involved healthcare provider. Group 1 (n=45) will receive bilateral sphenopalatine ganglion blocks with 4 mL of 0.5% bupivacaine applied intranasally using cotton-tipped applicators. Group 2 (n=45) will receive bilateral infraorbital nerve blocks with 4 mL of 0.5% bupivacaine under ultrasound guidance. Both blocks will be performed after anesthesia induction but before the start of surgery.

All patients will undergo standardized general anesthesia using propofol, fentanyl, and rocuronium for induction, followed by maintenance with remifentanil infusion and propofol titration to maintain BIS 40-60. Analgesic medications such as paracetamol, dexketoprofen, and dexamethasone will be administered intraoperatively. At the end of surgery, neuromuscular blockade will be reversed with sugammadex, and patients will be extubated when the TOF ratio exceeds 0.9.

Postoperative assessments include pain severity using the Visual Analog Scale (VAS), agitation level using the Richmond Agitation-Sedation Scale (RASS), and postoperative nausea and vomiting (PONV) using the Verbal Descriptive Scale (VDS). Rescue analgesia (morphine) and antiemetic (ondansetron) use will be recorded. The primary outcome is the quality of recovery measured by the QoR-15 questionnaire at 24 hours postoperatively. Secondary outcomes include intraoperative anesthetic consumption, total opioid requirement within 24 hours, time to first analgesic use, facial edema/hematoma, and PACU discharge time using the Modified Aldrete Score.

All interventions and assessments will be performed by blinded observers, and no placebo or experimental drugs will be used. No biological specimens will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Scheduled for elective septorhinoplasty under general anesthesia
* ASA physical status I-II
* Able to understand and sign informed consent

Exclusion Criteria:

* Local infection at the injection site
* History of psychiatric or neurological disorders that impair questionnaire response
* Known coagulopathy
* Allergy to local anesthetics
* History of chronic pain or use of chronic analgesic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery at postoperative 24 hours | 24 hours postoperatively
  Postoperative recovery will be assessed using the Quality of Recovery-15 (QoR-15) questionnaire. The scale contains 15 items covering pain, physical comfort, emotional state, physical independence, and psychological support. Each item is scored from 0 to 10, and the total score ranges from 0 to 150. Higher scores indicate better recovery.

SECONDARY OUTCOMES:
Pain severity over 24 hours | 1 to 24 hours postoperatively
  Postoperative pain intensity will be measured using the Visual Analog Scale (VAS) at 1, 2, 6, 12, and 24 hours. The scale ranges from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No